CLINICAL TRIAL: NCT02241655
Title: Electroencephalography Guidance of Anesthesia to Alleviate Geriatric Syndromes (ENGAGES) Study
Brief Title: Electroencephalography Guidance of Anesthesia
Acronym: ENGAGES
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Michael Avidan, Professor of Anesthesiology, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 201407128; 1UH2AG050312-01 (NIH)
Record Dates: First submitted 2014-09-11; First posted 2014-09-16 (Estimated); Results first posted 2019-06-18 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Delirium
Keywords: Anesthesia; Electroencephalography; Burst suppression; Surgery; Delirium; Falls; Health related quality of life
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EEG guided protocol (Experimental): Participants will have a pragmatic EEG-guided anesthetic protocol during their surgery. Practitioners will modify administration of anesthesia in an attempt to limit the occurrence of EEG burst suppression or persistent suppression.
  Interventions: Device: a pragmatic EEG-guided anesthetic protocol
- Control Arm (No Intervention): Participants will have the standard anesthetic protocol.

INTERVENTIONS:
Device: a pragmatic EEG-guided anesthetic protocol
  Other Names: Bispectral Index proprietary processed EEG monitor
  Arms: EEG guided protocol

SUMMARY:
This study aims to determine whether, compared with usual anesthetic care, an electroencephalography-guided anesthesia protocol is effective at preventing postoperative delirium and its downstream effects, and improving postoperative patient reported health-related quality of life.

DETAILED DESCRIPTION:
Delirium is one of several geriatric syndromes, and is among the most common postoperative complications, affecting up to 70% of surgical patients older than 60. Delirium is an acute change that manifests as inattention and inability to think logically, and is deeply distressing to patients and their families. Based on our surveys of 1,000 surgical patients, over 30% were worried about experiencing delirium. Delirious patients are unable to participate effectively in rehabilitation exercises and are susceptible to other geriatric syndromes, like falls. The occurrence and duration of delirium are associated with longer intensive care unit and hospital stay, persistent cognitive deterioration, hospital readmission and increased mortality rate. Additionally, delirium carries a huge social and economic burden, costing over $60,000 per patient per year. Despite the importance of delirium to patients and to society, no approach has been proven to prevent postoperative delirium. Furthermore postoperative delirium is frequently unrecognized, and surgical patients are not followed systematically after they are discharged from hospital. Without diagnosing delirium or following patients postoperatively, we are limited in our ability to test the effectiveness of any intervention to prevent or treat postoperative delirium and its sequelae. There is mounting evidence that electroencephalography guidance of general anesthesia can decrease postoperative delirium. Specifically, our group has found that a suppressed electroencephalogram pattern, which occurs with deep anesthesia, is associated with increased delirium and death after surgery. The Electroencephalography Guidance of Anesthesia to Alleviate Geriatric Syndromes (ENGAGES) Study will therefore compare the effectiveness of two anesthetic protocols for reduction of postoperative delirium. One protocol will be based on current standard anesthetic practice, and the other protocol will be based on electroencephalography guidance. We also expect to determine the impact of the anesthetic protocols on patient reported outcomes of health-related quality of life. At Washington University, we have successfully implemented an ambitious study that enrolls patients at the preoperative assessment clinic, and tracks their health and wellbeing at 30 days and at 1-year postoperatively. This will enable us to assess the consequences of postoperative delirium and to determine whether anesthetic management can impact patient reported outcomes, such as health-related quality of life. We shall also explore whether a multi-component safety intervention for delirious patients prevents downstream adverse events, like falls. The ENGAGES study - through its structured anesthesia protocols, its thorough approach to delirium assessment, and its ability to track patients' health and wellbeing postoperatively - is poised to make a major contribution to the care of elderly patients who are at risk of postoperative delirium and other adverse outcomes.

ELIGIBILITY:
Inclusion:

* Patients 60 years old and older,
* Competent to provide informed consent
* Undergoing major elective surgery that requires a minimum stay of 2 days postoperatively (e.g., open cardiac surgery, open thoracic surgery, major vascular surgery, intra-abdominal surgery, open gynecologic surgery, open urologic surgery, major orthopedic surgery, open hepato-biliary surgery and major ear, nose and throat surgery)

Exclusions

* Neurosurgical procedures will be excluded as surgery on the brain can confound the outcome (postoperative delirium).
* Patients with preoperative delirium and patients who are unable to participate adequately in delirium screening including those who are blind, deaf, or illiterate or fluent in languages other than English.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1400 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2020-10 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Michael S. Avidan, MBBCh, FCASA, Principal Investigator — Washington University School of Medicine; Eric Lenze, MD, Study Director — Washington University School of Medicine; Nan Lin, PhD, Study Director — Washington University School of Medicine; Susan Stark, PhD, Study Director — Washington University School of Medicine; Troy Wildes, MD, Study Director — Washington University School of Medicine; Anke Winter, MD, Study Director — Washington University School of Medicine; Sharon Inouye, MD, Study Director — Hebrew Rehabilitation Center; Arbi Ben Abdallah, PhD, Study Director — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Derived] Guay CS, Kafashan M, Huels ER, Jiang Y, Beyoglu B, Spencer JW, Geczi K, Apakama G, Ju YS, Wildes TS, Avidan MS, Palanca BJA. Postoperative Delirium Severity and Recovery Correlate With Electroencephalogram Spectral Features. Anesth Analg. 2023 Jan 1;136(1):140-151. doi: 10.1213/ANE.0000000000006075. Epub 2022 May 13. PMID 36130079
- [Derived] Fritz BA, King CR, Mickle AM, Wildes TS, Budelier TP, Oberhaus J, Park D, Maybrier HR, Ben Abdallah A, Kronzer A, McKinnon SL, Torres BA, Graetz TJ, Emmert DA, Palanca BJ, Stevens TW, Stark SL, Lenze EJ, Avidan MS; ENGAGES Research Group. Effect of electroencephalogram-guided anaesthesia administration on 1-yr mortality: follow-up of a randomised clinical trial. Br J Anaesth. 2021 Sep;127(3):386-395. doi: 10.1016/j.bja.2021.04.036. Epub 2021 Jul 7. PMID 34243940
- [Derived] Wildes TS, Mickle AM, Ben Abdallah A, Maybrier HR, Oberhaus J, Budelier TP, Kronzer A, McKinnon SL, Park D, Torres BA, Graetz TJ, Emmert DA, Palanca BJ, Goswami S, Jordan K, Lin N, Fritz BA, Stevens TW, Jacobsohn E, Schmitt EM, Inouye SK, Stark S, Lenze EJ, Avidan MS; ENGAGES Research Group. Effect of Electroencephalography-Guided Anesthetic Administration on Postoperative Delirium Among Older Adults Undergoing Major Surgery: The ENGAGES Randomized Clinical Trial. JAMA. 2019 Feb 5;321(5):473-483. doi: 10.1001/jama.2018.22005. PMID 30721296
- [Derived] Maybrier HR, King CR, Crawford AE, Mickle AM, Emmert DA, Wildes TS, Avidan MS, Palanca BJA; ENGAGES Study Investigators. Early Postoperative Actigraphy Poorly Predicts Hypoactive Delirium. J Clin Sleep Med. 2019 Jan 15;15(1):79-87. doi: 10.5664/jcsm.7576. PMID 30621829
- [Derived] Aranake-Chrisinger A, Cheng JZ, Muench MR, Tang R, Mickle A, Maybrier H, Lin N, Wildes T, Lenze E, Avidan MS. Ability of postoperative delirium to predict intermediate-term postoperative cognitive function in patients undergoing elective surgery at an academic medical centre: protocol for a prospective cohort study. BMJ Open. 2018 Mar 17;8(3):e017079. doi: 10.1136/bmjopen-2017-017079. PMID 29550773
- [Derived] Mickle AM, Maybrier HR, Winter AC, McKinnon SL, Torres BA, Lin N, Lenze EJ, Stark S, Muench MR, Jacobsohn E, Inouye SK, Avidan MS, Wildes TS; ENGAGES Research Group*. Achieving Milestones as a Prerequisite for Proceeding With a Clinical Trial. Anesth Analg. 2018 Jun;126(6):1851-1858. doi: 10.1213/ANE.0000000000002680. PMID 29239943
- [Derived] Cui V, Tedeschi CM, Kronzer VL, McKinnon SL, Avidan MS. Protocol for an observational study of delirium in the post-anaesthesia care unit (PACU) as a potential predictor of subsequent postoperative delirium. BMJ Open. 2017 Jul 10;7(7):e016402. doi: 10.1136/bmjopen-2017-016402. PMID 28698343
- [Derived] Wildes TS, Winter AC, Maybrier HR, Mickle AM, Lenze EJ, Stark S, Lin N, Inouye SK, Schmitt EM, McKinnon SL, Muench MR, Murphy MR, Upadhyayula RT, Fritz BA, Escallier KE, Apakama GP, Emmert DA, Graetz TJ, Stevens TW, Palanca BJ, Hueneke R, Melby S, Torres B, Leung JM, Jacobsohn E, Avidan MS. Protocol for the Electroencephalography Guidance of Anesthesia to Alleviate Geriatric Syndromes (ENGAGES) study: a pragmatic, randomised clinical trial. BMJ Open. 2016 Jun 15;6(6):e011505. doi: 10.1136/bmjopen-2016-011505. PMID 27311914

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1400 participants were consented to the study168 were not randomized to a study treatment arm (2 died, 49 were ineligible after enrollment, 49 surgery was cancelled, 31 research team missed the surgery, 37 withdrew). A total of 1232 patients were randomized to a study arm.
Groups:
- EEG Guided Protocol: Participants will have a pragmatic EEG-guided anesthetic protocol during their surgery. Practitioners will modify administration of anesthesia in an attempt to limit the occurrence of EEG burst suppression or persistent suppression.
  a pragmatic EEG-guided anesthetic protocol
Period: Overall Study
Arm/Group | EEG Guided Protocol | Control Arm
Started | 614 | 618
Completed | 614 | 618
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | EEG Guided Protocol | Control Arm | Total
Number analyzed (Participants) | 614 | 618 | 1232
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 69.5 [65.0 to 74.7] | 69.4 [64.7 to 75.8] | 69.5 [64.8 to 75.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 282 | 281 | 563
  Male | 332 | 337 | 669
Race/Ethnicity, Customized [Number; unit: participants]
  White | 555 | 558 | 1113
  Black | 54 | 53 | 107
  Other | 5 | 7 | 12
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 614 | 618 | 1232
BMI [Median (Inter-Quartile Range); unit: kg/m^2] | 29.0 [25.0 to 33.0] | 29.0 [25.0 to 33.0] | 29.0 [25.0 to 33.0]
Attended College [Count of Participants; unit: Participants] | 198 | 208 | 406
Lifetime tobacco use [Count of Participants; unit: Participants] | 376 | 349 | 725
Number of Participants with a Weekly Alcohol Intake [Count of Participants; unit: Participants] | 289 | 297 | 586
Current use of anticonvulsants [Count of Participants; unit: Participants] | 94 | 81 | 175
Regular use of opioids [Count of Participants; unit: Participants] | 154 | 149 | 303
Regular use of benzodiazepine [Count of Participants; unit: Participants] | 86 | 102 | 188
Number of participants with American Society of Anesthesiologist Classification greater than 3 [Count of Participants; unit: Participants] — American Society of Anesthesiologist (ASA) Classification ASA I: Normal Healthy patient ASA II: A patient with mild systemic disease ASA III: A patient with severe systemic disease ASA IV: a patient with severe systemic disease that is a constant threat to life ASA V: A moribund patient who is not expected to survive without the operation ASA VI: A declared brain-dead patient whose organs are being removed for donor purposes
  Participants | 209 | 221 | 430
Marginal exercise tolerance (METs) less than 4 [Count of Participants; unit: Participants] — The Functional status of the patient can be divided into POOR (< 4 METs,-unable to walk > 2 blocks on level ground without stopping due to symptoms, eating, dressing, toileting, walking indoors, light housework) or MODERATE /EXCELLENT (> 4 METs, -climbing > 1 flight of stairs without stopping, walking up hill > 1-2 blocks, scrubbing floors, moving furniture, golf, bowling, dancing or tennis, running short distance
  Participants | 297 | 295 | 592
Pulmonary hypertension [Count of Participants; unit: Participants] | 97 | 95 | 192
Aortic stenosis [Count of Participants; unit: Participants] | 90 | 108 | 198
History or high risk OSA [Count of Participants; unit: Participants] | 230 | 219 | 449
History of delirium [Count of Participants; unit: Participants] | 78 | 79 | 157
Number of comorbidities [Median (Inter-Quartile Range); unit: Number of comorbidities] | 5 [3 to 6] | 5 [3 to 6] | 5 [3 to 6]
History of depression [Count of Participants; unit: Participants] | 85 | 83 | 168
Personal Health Questionnaire Depression Scale (PHQ-8) [Median (Inter-Quartile Range); unit: units on a scale] — Assesses current depression. Range 0 to 24. greater than or equal to 10 indicates major depression and greater than or equal to 20 indicates severe major depression.
  units on a scale | 3 [1 to 6] | 3 [0 to 6] | 3.0 [0.0 to 6.0]
Short Blessed Test (SBT) [Median (Inter-Quartile Range); unit: units on a scale] — The SBT is a screening tool that aids in detecting early cognitive changes associated with dementia disorders. Rage 0 to 28. A score of 0-4 is normal cognition, 5-9 is questionable cognitive impairment, 10 or greater is cognitive impairment consistent with dementia.
  units on a scale | 2 [0 to 4] | 2 [0 to 4] | 2.0 [0.0 to 4.0]
8-item Inerview-Differentiate Aging and Dementia (AD8) [Median (Inter-Quartile Range); unit: units on a scale] — The AD8 is quite sensitive to detecting early cognitive changes associated many common dementing illness including Alzheimer disease, vascular dementia, Lewy body dementia and frontotemporal dementia. Range 0 to 8. A score of 0-1 is normal cognition, 2 or greater cognitive impairment is likely to be present.
  units on a scale | 0 [0 to 1] | 0 [0 to 1] | 0.0 [0.0 to 1.0]
Barthel Activies of Daily Living [Median (Full Range); unit: units on a scale] — Assesses functional independence. Range 0 to 100. Less than 20 indicates totally dependent, 20 to 39 indicates very dependent, 40-59 indicates partially dependent, 60 to 79 indicates minimally dependent, 80 to 100 indicates independent.
  units on a scale | 15 [15 to 15] | 15 [15 to 15] | 15 [15 to 15]
Hand grip strength [Mean (Standard Deviation); unit: kg] | 26.4 (11.0) | 25.7 (10.7) | 26.1 (10.9)
Timed up and go [Median (Inter-Quartile Range); unit: seconds] | 10.5 [9.2 to 13.1] | 11.0 [9.4 to 13.4] | 10.8 [9.3 to 13.2]
Lawton Instrumental Activities of Daily Living [Median (Inter-Quartile Range); unit: units on a scale] — Instrument assesses independent living skills. Range 0 (low function, dependent) to 8 (high function, independent).
  units on a scale | 8 [7 to 8] | 8 [8 to 8] | 8 [7 to 8]
Physical Veterans Rand 12 Item Health Survey (VR-12) Score [Mean (Standard Deviation); unit: Physical Score] — VR-12 is a patient reported global heath measure that is used to assess a patient's overall perspective of their health. Answers are summarized into two scores, a Physical Component Score and a Mental Component Score which then provides an important contrast between the respondents physical and psychological health status. Standardized scale 0 to 100 with 50 representing the population average. A score above 50 is better than the USA average where a score below 50 is worse than the USA average.
  Physical Score | 38.1 (11.9) | 38.2 (11.8) | 38.1 (11.8)
Mental VR-12 score [Mean (Standard Deviation); unit: Mental Score] — VR-12 is a patient reported global heath measure that is used to assess a patient's overall perspective of their health. Answers are summarized into two scores, a Physical Component Score and a Mental Component Score which then provides an important contrast between the respondents physical and psychological health status. Standardized scale 0 to 100 with 50 representing the population average. A score above 50 is better than the USA average where a score below 50 is worse than the USA average.
  Mental Score | 53.6 (10.6) | 53.6 (11.0) | 53.6 (10.8)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Delirium
Description: Delirium will be assessed at baseline and then once a day postoperative for up to 5 days. Patients were assessed for delirium using the Confusion Assessment Method for verbal patients or the Confusion Assessment Method for the Intensive Care Unit for non verbal or intubated patients, and patients medical records were reviewed for evidence of delirium by doctors and nurses assessments. Patients were considered to have delirium by any modality at anytime postoperative day one through five.
Time Frame: 5 days
Population: A total of 1232 patients were randomized (614 EEG guided protocol and 618 control arm). In the EEG guided group 10 patients could not be assessed for delirium (6 comatose, 2 withdrew, 2 early hospital discharge). In the control arm 9 patients could not be assessed for delirium (1 died, 5 comatose, 1 withdrew, 2 early hospital discharge).
Measure: Count of Participants; unit: Participants
Arm/Group | EEG Guided Protocol | Control Arm
Number analyzed (Participants) | 604 | 609
Participants | 157 | 140

2. Secondary Outcome: Postoperative Falls
Description: The hypothesis is that the EEG-guided anesthetic protocol and providing a safety intervention will prevent subsequent injurious falls. Falls will be assessed using the Prevention of Falls Network Europe (ProFaNE) questions. At baseline questions will be asked about preoperative falls, and at 30-days and 1-year postoperatively, questions will be asked about postoperative falls.
Time Frame: Up to 1 year postoperatively
Reporting Status: Not Posted, anticipated posting 2020-12

3. Secondary Outcome: Health Related Quality of Life
Description: The hypothesis is that the EEG-guided anesthetic protocol will improve postoperative quality of life. Patient self-reported Health-related Quality of Life information will be assessed through the Veteran's RAND 12-item Health Survey at baseline and during follow-up (30-day and 1-year).
Time Frame: Up to one year postoperatively
Reporting Status: Not Posted, anticipated posting 2020-12

4. Other Pre Specified Outcome: Duration of Delirium
Description: Duration will be calculated by the number of positive CAM,CAM-ICU or delirium chart reviews.
Time Frame: 5 days
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | EEG Guided Protocol | Control Arm
Number analyzed (Participants) | 604 | 609
days | 1 [1 to 3] | 1 [1 to 3]

5. Other Pre Specified Outcome: Agreements Among the FAM-CAM, Researchers' Delirium Assessments and Patient Perceptions
Description: The Family Confusion Assessment Method (FAM-CAM) instrument has previously been shown to have good agreement with the CAM and with DSM-IV diagnostic criteria in patients with cognitive impairment and in hospitalized patients.
Time Frame: 5 days
Reporting Status: Not Posted, anticipated posting 2020-07

6. Other Pre Specified Outcome: Duration or Recurrence of Delirium After Hospital Discharge
Description: As measured by the FAM-CAM and patient perceptions
Time Frame: 30 days post discharge
Reporting Status: Not Posted, anticipated posting 2020-07

7. Other Pre Specified Outcome: Clinically Relevant Outcomes Associated With Delirium
Description: Delirium incidence, duration and severity have all been shown to be associated with other (downstream) clinically relevant outcomes, including mortality, length of ICU stay, length of hospital stay, falls, cognitive decline and functional decline.
Time Frame: 1 year
Reporting Status: Not Posted, anticipated posting 2020-12

8. Other Pre Specified Outcome: Comparison of Patient-reported and Observational Pain Scores
Description: Given that postoperative delirium is common and may relate to uncontrolled pain, this has important implications for the assessment and treatment of postoperative pain. We plan to compare patient reported and behavioral pain assessments in both non-delirious and delirious patients.
Time Frame: 5 days
Reporting Status: Not Posted, anticipated posting 2020-07

9. Other Pre Specified Outcome: Postoperative Actigraphy
Description: Postoperative disturbances in sleep abnormalities have previously been associated with postoperative delirium. Measures of root mean-squared activity (RMSactivity) was calculated by combining counts (binned in 1-minute intervals) across all three accelerometer axes (X, Y, and Z) from 16:00 on the day of surgery to 6:00 the following day. Median activity count was calculated from all minutes with nonzero RMS activity within each epoch- higher values indicate more movement.
Time Frame: 1 day
Population: A total of 84 patients had analyzable data and included in the analysis. Patients were pooled regardless of intervention (EEG guidance or usual care) since the primary outcome was to assess whether using actigraphy could predict delirium regardless of interventions. Therefore, patients were separated by delirious and non-delirious patients.
Measure: Median (Inter-Quartile Range); unit: minutes RMSactivity>0
Groups:
- No Delirium: intact with no delirium throughout postoperative days (POD) 0-5
- Delirium POD 0-1: Patients who were delirious POD 0-1
- Delirium POD 2-5: Patients who were delirious POD 2-5
Arm/Group | No Delirium | Delirium POD 0-1 | Delirium POD 2-5
Number analyzed (Participants) | 51 | 24 | 13
minutes RMSactivity>0 | 134 [59 to 195] | 101 [50 to 141] | 93 [36 to 236]

10. Other Pre Specified Outcome: Relationship Between Clinical CAM-ICU and Rigorous Delirium Assessments
Description: Routine clinical (i.e. conducted by ICU nursing staff) delirium assessments in the intensive care units (conducted with the CAM-ICU) will be collected when these are available. Comparison will be made on the outcome of the assessment (positive for delirium or negative by delirium) between these routine clinical assessments and the assessments made by the research team. Since the purpose of this is to determine whether clinical staff are picking up episodes of delirium compared to researcher's assessment in all patients regardless of treatment group, data from both treatment arms were combined for the analysis.
Time Frame: 5 days
Population: Patients who were in the ICU, had a nursing CAM-ICU assessment and researcher's delirium assessment were included in this analysis. Agreement between the instruments was calculated using Kappa agreement.
Measure: Number (95% Confidence Interval); unit: Cohen's kappa coefficient
Groups:
- Patients With Nursing ICU Assessment: Patients who were in the ICU and had a nursing CAM-ICU and researcher's delirium assessment were included in this analysis.
Arm/Group | Patients With Nursing ICU Assessment
Number analyzed (Participants) | 562
Cohen's kappa coefficient | 0.37 [0.29 to 0.44]

11. Other Pre Specified Outcome: Postoperative Outcomes Hypothesized to be Associated With Anesthetic Depth
Description: There is an ongoing randomized, clinical trial investigating the effects of depth of anesthesia on a range of outcomes98, including death, myocardial infarction, cardiac arrest, pulmonary embolus, stroke, surgical site infection, ICU length of stay, hospital length of stay, intraoperative awareness, persistent pain and cancer recurrence. Many of these outcomes are tracked with the SATISFY-SOS study, and will therefore be reported for patients enrolled in the ENGAGES study.
Time Frame: 1 year
Reporting Status: Not Posted, anticipated posting 2020-12

12. Other Pre Specified Outcome: Delirium Prediction Models
Description: It is important to improve our understanding of factors that are associated with an increased incidence of postoperative delirium or perhaps may even mediate an elevated risk for postoperative delirium. The arm/group was included in the model to determine if it was associated with postoperative delirium therefore data is not presented by arm/group.
Time Frame: 5 days
Population: Covariated included were pre-selected and considered likely to be associated with postoperative delirium.
Measure: Number (95% Confidence Interval); unit: odds ratio
Groups:
- Regression Analysis: The purpose of the logistic regression and adjustment for prognostic covariates was to improve the power of the trial to detect a beneficial effect attributable to the intervention (minimization of electroencephalographic suppression) or to usual anesthesia care on the outcome of interest, postoperative delirium.
Arm/Group | Regression Analysis
Number analyzed (Participants) | 1051
odds ratio
  Guided Group | 1.12 [0.30 to 1.64]
  Age | 1.04 [1.02 to 1.06]
  Male | 0.99 [0.71 to 1.38]
  White | 0.46 [0.28 to 0.74]
  Living alone | 0.91 [0.63 to 1.32]
  Hearing aid use | 0.82 [0.52 to 1.30]
  No. Comorbidities | 1.08 [1.01 to 1.16]
  ASA greater than 3 | 1.98 [1.27 to 3.09]
  Marginal exercise tolerance less than 4 METS | 1.21 [0.86 to 1.70]
  Falls in previous 6 months | 1.25 [0.88 to 1.76]
  History of delirium | 1.83 [1.21 to 2.76]
  Preoperative PHQ8 | 1.03 [0.99 to 1.07]
  Preoperative Lawton | 0.95 [0.83 to 1.09]
  Preoperative Barthel | 0.95 [0.81 to 1.12]
  Preoperative opioids | 1.27 [0.88 to 1.82]
  Preoperative benzodiazepines | 1.28 [0.85 to 1.94]
  Preoperative sodium level | 0.98 [0.94 to 1.03]
  Preoperative creatinine level | 1.06 [0.91 to 1.22]
  Preoperative hemoglobin level | 0.99 [0.91 to 1.08]
  Cardiac surgery | 0.92 [0.58 to 1.44]

13. Other Pre Specified Outcome: Collaborations With Other Studies
Description: The ENGAGES study is being conducted in collaboration with complementary trials at the University of California, San Francisco (UCSF) (NCT01983384), the University of Michigan in Ann Arbor and the University of Manitoba in Winnipeg. Some of the outcomes will be analyzed considering data from some or all of these studies, as appropriate. In terms of the practicality of disseminating the EEG-guided protocol in North America and beyond, it will be important to demonstrate the feasibility and impact of the protocol in multiple sites.
Time Frame: 5 years
Reporting Status: Not Posted, anticipated posting 2025-01

14. Other Pre Specified Outcome: Number of Participants With Severe Delirium
Description: The severity of delirium will be scored using the CAM-Severity (CAM-S) metric, which has specifically been shown to be strongly associated with clinically relevant outcomes. Severe delirium was defined as patients with a CAM-S score of 10 or greater (range 0-19).
Time Frame: 5 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | EEG Guided Protocol | Control Arm
Number analyzed (Participants) | 604 | 609
Participants | 59 | 51

15. Other Pre Specified Outcome: EEG and Delirium
Description: EEG abnormalities have previously been associated with postoperative delirium
Time Frame: 5 days
Reporting Status: Not Posted, anticipated posting 2020-07

16. Other Pre Specified Outcome: Postoperative Actigraphy- Immobile Minutes
Description: Postoperative disturbances in sleep abnormalities have previously been associated with postoperative delirium. Measures of root mean-squared activity (RMSactivity) was calculated by combining counts (binned in 1-minute intervals) across all three accelerometer axes (X, Y, and Z) from 16:00 on the day of surgery to 6:00 the following day. We quantified inactivity using the number of immobile minutes, defined as the total number of minutes with an RMSactivity count of zero- higher number indicates patient had more time being immobile.
Time Frame: 1 day
Population: as for outcome 9
Measure: Median (Inter-Quartile Range); unit: minutes RMSactivity=0
Arm/Group | No Delirium | Delirium POD 0-1 | Delirium POD 2-5
Number analyzed (Participants) | 51 | 24 | 13
minutes RMSactivity=0 | 548 [472 to 625] | 584 [430 to 620] | 604 [440 to 683]

ADVERSE EVENTS:
Time Frame: Adverse events were collected during surgery up to 30 days postoperatively
Arm/Group | EEG Guided Protocol | Control Arm
All-Cause Mortality (participants affected / at risk) | 4/614 | 20/618
Serious Adverse Events (participants affected / at risk) | 124/614 | 130/618
Other Adverse Events (participants affected / at risk) | 361/614 | 345/618
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | EEG Guided Protocol (N=614) | Control Arm (N=618)
Bleeding/anemia requiring unexpected transfusion (Blood and lymphatic system disorders) | 5 | 11
Embolus (Blood and lymphatic system disorders) | 1 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1
Thrombosis without embolus (Blood and lymphatic system disorders) | 1 | 5
Other hematologic event (Blood and lymphatic system disorders) | 1 | 0
Cardiac Arrest (Cardiac disorders) | 1 | 12
Cardiac tamponade (Cardiac disorders) | 1 | 0
Congestive heart failure (Cardiac disorders) | 4 | 2
Myocardial infarction (Cardiac disorders) | 3 | 5
Unexpected atrial fibrillation (Cardiac disorders) | 2 | 2
Unexpected cardiogenic shock (Cardiac disorders) | 2 | 6
Unexpected heart block (Cardiac disorders) | 3 | 3
Other unexpected abnormal heart rhythms (Cardiac disorders) | 0 | 5
Unexpected hypo or hyperkelemia (Endocrine disorders) | 1 | 0
Unexpected hypo or hypernatremia (Endocrine disorders) | 0 | 1
Other endocrine or metabolic event (Endocrine disorders) | 3 | 5
Anastomotic leak (Gastrointestinal disorders) | 0 | 3
Nausea and/or vomiting (Gastrointestinal disorders) | 8 | 3
GI bleed (Gastrointestinal disorders) | 5 | 1
Ileus/bowel obstruction (Gastrointestinal disorders) | 12 | 8
Other GI event (Gastrointestinal disorders) | 14 | 18
Anaphylaxis (Immune system disorders) | 2 | 1
Infectious colitis (Immune system disorders) | 1 | 4
Sepsis (Immune system disorders) | 9 | 11
UTI (Immune system disorders) | 2 | 1
Wound infection (Immune system disorders) | 11 | 13
Other immune or infectious event (Immune system disorders) | 1 | 3
Anoxic encephalopathy (Nervous system disorders) | 0 | 1
Stroke (Nervous system disorders) | 10 | 4
Pain (Nervous system disorders) | 2 | 0
Other neurological event (Nervous system disorders) | 3 | 4
Hemothorax (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 10 | 3
pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory Failures (Respiratory, thoracic and mediastinal disorders) | 21 | 27
Other respiratory event (Respiratory, thoracic and mediastinal disorders) | 6 | 2
Acute kidney injury (Renal and urinary disorders) | 1 | 6
Renal failure requiring dialysis (Renal and urinary disorders) | 6 | 7
Urinary retention (Renal and urinary disorders) | 1 | 0
Other renal event (Renal and urinary disorders) | 3 | 3
Non-cardiogenic shock (Vascular disorders) | 4 | 1
Unexpected hypotension (Vascular disorders) | 4 | 1
Other vascular event (Vascular disorders) | 7 | 9
Other body system event (Surgical and medical procedures) | 12 | 14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | EEG Guided Protocol (N=614) | Control Arm (N=618)
Bleeding/anemia requiring unexpected transfusion (Blood and lymphatic system disorders) | 121 | 126
Embolus (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 24 | 23
Thrombosis without embolus (Blood and lymphatic system disorders) | 15 | 12
Other hematologic event (Blood and lymphatic system disorders) | 2 | 1
Myocardial infarction (Cardiac disorders) | 0 | 5
Unexpected atrial fibrillation (Cardiac disorders) | 73 | 97
Unexpected cardiogenic shock (Cardiac disorders) | 6 | 5
Unexpected heart block (Cardiac disorders) | 17 | 15
Other unexpected abnormal heart rhythms (Cardiac disorders) | 9 | 15
Other cardiac event (Cardiac disorders) | 10 | 7
unexpected hypo or hyperglycemia (Endocrine disorders) | 0 | 5
Unexpected hypo or hyperkalemia (Endocrine disorders) | 9 | 3
Unexpected hypo or hypernatremia (Endocrine disorders) | 13 | 6
Other endocrine event (Endocrine disorders) | 5 | 5
Nausea and/or vomiting (Gastrointestinal disorders) | 9 | 10
GI bleed (Gastrointestinal disorders) | 2 | 3
Ileus/bowel obstruction (Gastrointestinal disorders) | 22 | 22
Other GI event (Gastrointestinal disorders) | 12 | 11
Infectious colitis (Immune system disorders) | 6 | 3
Non-anaphylactic allergic reaction (Immune system disorders) | 3 | 1
Sepsis (Immune system disorders) | 0 | 3
UTI (Immune system disorders) | 20 | 19
Wound infection (Immune system disorders) | 14 | 10
Other immune event (Immune system disorders) | 19 | 14
Stroke (Nervous system disorders) | 1 | 0
Pain (Nervous system disorders) | 4 | 1
Other neurological event (Nervous system disorders) | 7 | 8
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Hemothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Hypoxemia (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 11
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 6 | 10
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Respiratory Failures (Respiratory, thoracic and mediastinal disorders) | 9 | 10
Other respiratory event (Respiratory, thoracic and mediastinal disorders) | 24 | 17
Acute kidney injury (Renal and urinary disorders) | 40 | 40
Renal failure requiring dialysis (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 36 | 28
Other renal event (Renal and urinary disorders) | 20 | 20
Non-cardiogenic shock (Cardiac disorders) | 4 | 3
Unexpected hypertension (Vascular disorders) | 2 | 1
Unexpected hypotension (Vascular disorders) | 15 | 19
Other vascular event (Vascular disorders) | 8 | 11
Other body system event (Surgical and medical procedures) | 13 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan: Study protocol with analysis plan (2015-12-21): https://cdn.clinicaltrials.gov/large-docs/55/NCT02241655/Prot_SAP_001.pdf
  • Statistical Analysis Plan: Updated Analysis plan for 1 year (2019-06-21): https://cdn.clinicaltrials.gov/large-docs/55/NCT02241655/SAP_002.pdf